CLINICAL TRIAL: NCT01463306
Title: A 12-MONTH OPEN-LABEL STUDY TO EVALUATE THE SAFETY AND TOLERABILITY OF PREGABALIN AS ADJUNCTIVE THERAPY IN PEDIATRIC SUBJECTS 1 MONTH TO 16 YEARS OF AGE WITH PARTIAL ONSET SEIZURES AND PEDIATRIC AND ADULT SUBJECTS 5 TO 65 YEARS OF AGE WITH PRIMARY GENERALIZED TONIC-CLONIC SEIZURES
Brief Title: A 12-Month Study To Evaluate The Safety And Tolerability Of Pregabalin As Add-On Therapy In Pediatric Subjects 1 Month To 16 Years Of Age With Partial Onset Seizures And Pediatric And Adult Subjects 5 To 65 Years Of Age With Primary Generalized Tonic-Clonic Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Not Applicable | Masking: None | Purpose: Treatment
Other Study IDs: A0081106; 2011-001412-65 (EudraCT Number)
Record Dates: First submitted 2011-10-17; First posted 2011-11-01 (Estimated); Results first posted 2020-02-21 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2020-01

CONDITIONS: Epilepsy, Partial Seizures; Epilepsy, Primary Generalized Tonic-Clonic Seizures
Keywords: safety; partial onset seizures; primary generalized tonic-clonic seizures; pregabalin; pediatric; adult; open-label; long term
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open (Experimental): Pregabalin open label flexible dose
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — Pregabalin administered as either capsule or liquid oral formulations. Subjects <4 years of age at Visit 1 will receive study medication 3 times daily (TID) in equally divided doses. Subjects who are ≥4 years of age at Visit 1 will receive study medication twice daily (BID) in equally divided doses. Children less than 17 years of age will receive from 2.5 mg/kg/day to 10.0 mg/kg/day (maximum 600 mg/day. Adults 17 and older will receive from 150 mg/day to 600 mg/day.
  Other Names: Lyrica

SUMMARY:
Study A0081106 is a 12-month open-label study to evaluate the long term safety and tolerability of pregabalin as add-on therapy in pediatric subjects 1 month to 16 years of age with partial onset seizures and pediatric and adult subjects 5 to 65 years of age with primary generalized tonic-clonic seizures. Pregabalin will be administered in equally divided daily doses for 1 year, in either capsule or liquid oral formulation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects and/or parent(s)/legally acceptable representative must be considered willing and able to sign consent, and complete daily dosing and seizure diaries and complete all scheduled visits.
* Male and female epilepsy subjects, 1 month to 65 years of age inclusive on the date of the Screening Visit.
* Diagnosis of epilepsy with seizures classified as simple partial, complex partial, or partial becoming secondarily generalized, or primary generalized tonic-clonic seizures according to the International League Against Epilepsy (ILAE 2010) Diagnosis Criteria.
* Partial onset seizure subjects must have had an average of at least 3 seizures per 28 day period in the 3 months prior to screening.
* Currently receiving a stable dose of 1 to 3 antiepileptic drugs (stable within 28 days prior to screening).

Exclusion Criteria:

* Lennox-Gastaut syndrome, Infantile Spasms, Absence seizures, BECT (Benign Epilepsy with Centrotemporal Spikes), and Dravet syndrome,
* A current diagnosis of febrile seizures or any febrile seizure within 1 year of screening.
* Status epilepticus within 1 year prior to visit 1.
* Seizures related to drugs, alcohol, or acute medical illness.
* Progressive structural CNS lesion or a progressive encephalopathy.

Ages: 1 Month to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 605 (Actual)
Dates: Start 2012-02-21 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2019-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (147):
- United States (21):
  - Center for Neurosciences, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital Los Angeles, Los Angeles, California
  - Axcess Medical Research, Loxahatchee Groves, Florida
  - Laszlo J. Mate, M.D., P.A., North Palm Beach, Florida
  - Pediatric Epilepsy Center Of Central Florida, Orlando, Florida
  - Pediatric Neurology, PA, Orlando, Florida
  - Tallahassee Neurological Clinic, Tallahassee, Florida
  - Pediatric Epilepsy and Neurology Specialists, PA, Tampa, Florida
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Josephson Wallack Munshower Neurology P.C., Indianapolis, Indiana
  - Kosair Children's Hospital, Louisville, Kentucky
  - University of Louisville Physicians, Louisville, Kentucky
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Akron Children's Hospital, Akron, Ohio
  - Ohio Clinical Research Partners, LLC, Canton, Ohio
  - The children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Dallas Pediatric Neurology Associates, Dallas, Texas
  - Road Runner Research, Ltd., San Antonio, Texas
  - Rainier Clinical Research Center, Inc., Renton, Washington
- Belarus (2):
  - GU Republican Scientific and Practical Center Mother and Child, Minsk
  - UZ Vitebsk Regional Childrens Clinical Centre, Vitebsk
- Belgium (3):
  - Hopital Universitaire Des Enfants Reine Fabiola, Brussels, Brussels Capital
  - Hospital Erasme, Brussels, Brussels Capital
  - UZ Brussel - Campus Jette - Pediatric Neurology, Brussels, Brussels Capital
- Bosnia and Herzegovina (3):
  - University Clinical Center Sarajevo, Sarajevo, Canton Sarajevo, Bosnia and Herzegovina
  - University Clinical Hospital Mostar, Mostar, Herzegovina-neretva Canton
  - Public Health Institution Hospital "Dr. Mladen Stojanovic", Prijedor, Republika Srpska
- Bulgaria (6):
  - "Multiprofile Hospital for Active Treatment Puls" AD, Blagoevgrad
  - UMHAT Dr. Georgi Stranski Ltd., Pleven
  - MHAT Central Onco Hospital OOD, Plovdiv
  - UMHAT "Sveti Georgi" Ltd., Pediatric Clinic, Plovdiv
  - MHATNP Sveti Naum EAD, Sofia
  - DCC Sveta Anna - Sofia\ Neurological room, Sofia
- China (3):
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Shanghai Huashan Hospital, Shanghai, Shanghai Municipality
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
- Czechia (2):
  - Fakultni nemocnice Brno - Detska nemocnice, Brno - Cerna Pole
  - Fakultni nemocnice v Motole, Prague
- France (3):
  - Hopital Raymond Poincare, Garches
  - CHRU de Rennes - Hopital Pontchaillou, Rennes
  - Hopitaux Universitaire de Strasbourg - Hopital Hautepierre, Strasbourg
- Universitaetsklinikum Jena, Jena, Thuringia, Germany
- Greece (2):
  - General Children's Hospital of Athens "P&A Kyriakou", Athens
  - General Children's Hospital Penteli, Athens
- Hungary (8):
  - Dr. Kenessey Albert Kórház és Rendelőintézet, Balassagyarmat
  - Semmelweis Egyetem, I. Sz. Gyermekgyogyaszati Klinika/, Budapest
  - Szent Janos Korhaz es Eszak-budai Egyesitett Korhazak, Budapest
  - Szent Margit Korhaz, Budapest
  - Heim Pal Gyermekkorhaz, Neurologiai Osztaly, Budapest
  - Magyarorszagi Reformatus Egyhaz Bethesda Gyermekkorhaz, Gyermekneurologia, Budapest
  - Pest Megyei Flor Ferenc Korhaz, Neurologiai Osztaly, Kistarcsa
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
- India (3):
  - Mangala Hospital & Mangala Kidney Foundation, Mangalore, Karnataka
  - Getwell Hospital and Research Institute, Dhantoli, Nagpur, Maharashtra
  - KEM Hospital Research Centre, Pune, Maharashtra
- Israel (3):
  - Bnai Zion Medical Center, Haifa
  - Pharmacy of Tel Aviv Sourasky Medical Center, Tel Aviv
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (4):
  - A.O.U. Ospedali Riuniti di Ancona - Presidio Ospedaliero G. Salesi - S.O.D. Farmacia, Ancona
  - A.O.U. Ospedali Riuniti di Ancona Presidio Ospedaliero G. Salesi, Ancona
  - Azienda Ospedaliero-Universitaria Meyer, Florence
  - Fondazione Istituto Neurologico Nazionale Casimiro Mondino, IRCCS, Pavia
- Lebanon (2):
  - American University of Beirut Medical Center, Beirut
  - Saint George Hospital - University Medical Center, Beirut
- Malaysia (3):
  - Hospital Raja Perempuan Zainab II, Kota Bharu, Kelantan
  - Hospital Raja Permaisuri Bainun, Ipoh, Perak
  - Hospital Kuala Lumpur, Kuala Lumpur
- Pzu Neuron, Bijelo Polje, Montenegro
- Philippines (8):
  - Cebu Doctors' University Hospital, Cebu City, CEBU
  - Perpetual Succour Hospital, Cebu City
  - Philippine Children's Medical Center, Diliman, Quezon City
  - Manila Doctors Hospital, Manila
  - Metropolitan Medical Center, Manila
  - University of Santo Tomas Hospital, Manila
  - Capitol Medical Center Inc., Quezon City
  - St. Luke's Medical Center, Quezon City
- Poland (10):
  - COPERNICUS Podmiot Leczniczy Sp z o.o., Gdansk
  - Klinika Neurologii Rozwojowej, Gdansk
  - NZOZ Wielospecjalistyczna Poradnia Lekarska SYNAPSIS, Lech Szczechowski, Katowice
  - Nzoz Novo Med, Katowice
  - Gabinet lekarski Neurologii I Leczenia padaczki, Kielce
  - Niepubliczny Zaklad Opieki Zdrowotnej "HIPOKRATES-II" Sp. z o.o., Krakow
  - Instytut Medycyny Wsi im. Witolda Chodzki w Lublinie, Lublin
  - Katedra i Klinika Neurologii Wieku Rozwojowego, Poznan
  - NZOZ "IGNIS" Dr. n. med. Alicja Lobinska, Świdnik
  - Oddzial Neurologii Dzieciecej, Dolnoslaski Szpital Specjalistyczny im.T. Marciniaka,, Wroclaw
- Romania (5):
  - Spitalul clinic de copii Dr. Victor Gomoiu, Bucharest
  - Spitalul Clinic de Psihiatrie "Prof. Dr. Al. Obregia", Bucharest
  - Spitalul Clinic de Urgente pentru Copii "Sf. Maria", Iași
  - Spitalul de Psihiatrie Dr. Ghe. Preda, Sibiu
  - Centrul Medical Dr. Bacos Cosma, Timișoara
- Russia (16):
  - SPHI Leningrad Regional Psychoneurological Dispensary, Pgt. Roshchino, Leningradskaya Oblast'
  - Nizhmedklinika, Nizhny Novgorod, Nizhny Novgorod Oblast
  - Perm State Medical University n. a. acad. E.A. Vagner, Perm, Permskiy KRAY
  - State Budgetary Healthcare Institution of Stavropol region, Pyatigorsk, Stavropol Kray
  - TSBHI City Hospital No. 5 of Barnaul, Barnaul
  - FSFEI HE N.I. Pirogov RNRMU of Minzdrav of Russia, Moscow
  - Non-state Healthcare Institution, Moscow
  - Perm State Medical University n. a. acad. E.A. Vagner, Perm
  - LLC Medical Technologies, Saint Petersburg
  - SPHI Leningrad Regional Psychoneurological Dispensary, Saint Petersburg
  - FSBI V.M. Bekhterev National Research Medical Center, Saint Petersburg
  - SBHI of Saint Petersburg Psychoneurological Dispensary #5, Saint Petersburg
  - Regional State Budgetary Institution of Ministry of Health, Smolensk
  - RSBHI Smolensk Regional Clinical Hospital, Smolensk
  - GBOU VPO "Smolensk State Medical University", Smolensk
  - MAI Children's City Clinical Hospital No 9, Yekaterinburg
- Serbia (4):
  - Institute for Child and Youth Healthcare of Vojvodina, Novi Sad, Vojvodina
  - Mother and Child Healthcare Institute Dr Vukan Cupic, Belgrade
  - University Children's Hospital Belgrade, Belgrade
  - Clinical Center of Kragujevac, Kragujevac
- Singapore (2):
  - National University Hospital, Singapore
  - KK Women's and Children's Hospital, Singapore
- Neurologicka ambulancia MUDr. Eva Gasparova, Hlohovec, Slovakia
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Hospital Universitario Miguel Servet, Zaragoza, Spain
- Taiwan (3):
  - Chang Gung Memorial Hospital (CGMH) - Kaohsiung Branch, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- Thailand (2):
  - Siriraj Hospital, Mahidol University, Faculty of Medicine, Bangkoknoi, Bangkok
  - Phramongkutklao Hospital, Neurology Unit,, Ratchathevee, Bangkok
- Turkey (Türkiye) (7):
  - Hacettepe University Medical Faculty, Ankara, Ankara/sihhiye
  - Ege University Medical Faculty Department of Pediatrics Health and Diseases,, Izmir, Bornova/izmir
  - Karadeniz Technical University Faculty of Medicine Farabi Hospital, Trabzon, Farabi
  - Izmir Tepecik Training and Research Hospital, Izmir, Konak Turkey
  - Behcet Uz Children Disease and Surgery Training and Research Hospital, Izmir, Konak
  - Eskisehir Osmangazi University Medical Faculty, Eskişehir, Meselik Campus
  - Dokuz Eylül University medical Faculty Internal Medicine Disease, Izmir
- Ukraine (13):
  - Komunalnyi zaklad "Dnipropetrovska dytiacha miska klinichna likarnia #5", Dnipro
  - Komunalnyi zaklad "Dnipropetrovska oblasna dytiacha klinichna likarnia", Dnipropetrovsk
  - Ivano-Frankivska oblasna dytiacha klinichna likarnia, Ivano-Frankivsk
  - Derzhavna ustanova "Instytut nevrolohii, psykhiatrii ta narkolohii, Kharkiv
  - Komunalne nekomertsiine pidpryiemstvo Kharkivskoi oblasnoi rady "Oblasna klinichna psykhiatrychna li, Kharkiv
  - Derzhavnyi zaklad "Ukrainskyi medychnyi tsentr reabilitatsii ditei z orhanichnym urazhenniam, Kyiv
  - Komunalne nekomertsiine pidpryiemstvo Lvivskoi oblasnoi rady Lvivska oblasna klinichna likarnia, Lv, Lviv
  - Komunalna ustanova "Odeskyi oblasnyi medychnyi tsentr psykhichnoho zdorovia", Odesa
  - Komunalne nekomertsiine pidpryiemstvo "Odeskyi oblasnyi medychnyi tsentr psykhichnoho zdoroviaa", Odesa
  - KU "Odeska oblasna dytiacha klinichna likarnia", Odesa
  - Komunalna ustanova "Odeska oblasna psykhiatrychna likarnia No2", S. Oleksandrivka, Kominternivskyi R-n, Odeska Obl.
  - Oblasnyi klinichnyi tsentr neirokhirurhii ta nevrolohii, viddilennia neirokhirurhii No2, Uzhhorod
  - Komunalna ustanova "Miska klinichna likarnia #2", nevrolohichne viddilennia, Zaporizhzhia
- United Kingdom (2):
  - The Barberry National Centre for Mental Health, Birmingham, WEST Midlands
  - Salford Royal NHS Foundation Trust, Salford

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pility%20Of%20Pregabages/landing.aspx?StudyID=A0081106

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Reporting arms are on basis of pediatric and adult participants who consented to continue from previous studies receiving either pregabalin or placebo and pediatric participants who directly enrolled in this study. Previous studies- A0081041 (NCT01389596), A0081042 (NCT02072824), A0081105 (NCT01747915).
Groups:
- Pregabalin: Previous and Current: Pediatric and adult participants with partial onset seizures (POS) and primary generalized tonic-clonic (PGTC) seizures included in this arm are those who received pregabalin in previous studies. Pregabalin was administered in 3 equally divided doses per day (TID) when age less than (<) 4 years and in 2 equally divided doses per day (BID) when age greater than or equal to (>=) 4 years. Pediatric participants with body weight >=30 kilogram (kg) received pregabalin 2.5 milligram per kilogram per day (mg/kg/day) as liquid oral solution/capsule up to maximum of 10.0 mg/kg/day and with body weight <30 kg received pregabalin 3.5 mg/kg/day as liquid oral solution up to maximum of 14.0 mg/kg/day. Adult participants received pregabalin 150 milligram per day (mg/day) as liquid oral solution/oral capsule up to maximum of 600 mg/day. Maximum duration for treatment was 12 months.
- Placebo-Previous to Pregabalin-Current: Pediatric and adult participants with POS and PGTC seizures included in this arm are those who received placebo in previous studies. Pregabalin was administered TID when age <4 years and BID when age >= 4 years. Pediatric participants with body weight >=30 kg received pregabalin 2.5 mg/kg/day as liquid oral solution/capsule up to maximum of 10.0 mg/kg/day and with body weight <30 kg received pregabalin 3.5 mg/kg/day as liquid oral solution up to maximum of 14.0 mg/kg/day. Adult participants received pregabalin 150 mg/day as liquid oral solution/capsule up to maximum of 600 mg/day. Maximum duration for treatment was 12 months.
- Direct Pregabalin: Only pediatric participants with POS were enrolled in this arm who did not participate in any study previously. Pregabalin was administered TID when age <4 years and BID when age >= 4 years. Pediatric participants with body weight >=30 kg received pregabalin 2.5 mg/kg/day as liquid oral solution/capsule up to maximum of 10.0 mg/kg/day and with body weight <30 kg received pregabalin 3.5 mg/kg/day as liquid oral solution up to maximum of 14.0 mg/kg/day. Maximum duration for treatment was 12 months.
Period: Overall Study
Arm/Group | Pregabalin: Previous and Current | Placebo-Previous to Pregabalin-Current | Direct Pregabalin
Started | 384 | 210 | 11
Completed | 298 | 158 | 6
Not Completed | 86 | 52 | 5
Not completed — Adverse Event | 6 | 9 | 3
Not completed — Death | 3 | 3 | 0
Not completed — Lack of Efficacy | 22 | 16 | 1
Not completed — Lost to Follow-up | 5 | 2 | 0
Not completed — Protocol Violation | 4 | 0 | 0
Not completed — Withdrawal by Subject | 19 | 9 | 1
Not completed — Other | 26 | 13 | 0
Not completed — Approval expiry at site | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included participants who took at least 1 dose of the study medication in the study.
Groups:
- Pregabalin: Previous and Current: Pediatric and adult participants with POS and PGTC seizures included in this arm are those who received pregabalin in previous studies. Pregabalin was administered TID when age <4 years and BID when age >=4 years. Pediatric participants with body weight >=30 kg received pregabalin 2.5 mg/kg/day as liquid oral solution/capsule up to maximum of 10.0 mg/kg/day and with body weight <30 kg received pregabalin 3.5 mg/kg/day as liquid oral solution up to maximum of 14.0 mg/kg/day. Adult participants received pregabalin 150 mg/day as liquid oral solution/capsule up to maximum of 600 mg/day. Maximum duration for treatment was 12 months.
- Total: Total of all reporting groups
Arm/Group | Pregabalin: Previous and Current | Placebo-Previous to Pregabalin-Current | Direct Pregabalin | Total
Number analyzed (Participants) | 384 | 210 | 11 | 605
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.56 (11.43) | 13.03 (12.39) | 11.80 (3.87) | 12.71 (11.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 176 | 103 | 7 | 286
  Male | 208 | 107 | 4 | 319
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 85 | 47 | 1 | 133
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 0 | 4
  White | 294 | 160 | 9 | 463
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs), Treatment Emergent Serious Adverse Events (SAEs), Treatment Related AEs and Treatment Related SAEs
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment emergent are events between first dose of study drug and up to 28 days after last dose of study drug (up to 13 months) that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious AEs. Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Relatedness to study drug was assessed by the investigator.
Time Frame: Baseline (Day 1) up to 13 Months
Population: Safety population included participants who took at least 1 dose of the study medication in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin: Previous and Current | Placebo-Previous to Pregabalin-Current | Direct Pregabalin
Number analyzed (Participants) | 384 | 210 | 11
Participants
  Participants With AEs | 252 | 140 | 10
  Participants With SAEs | 53 | 23 | 1
  Participants With Treatment Related AEs | 104 | 65 | 9
  Participants With Treatment Related SAEs | 0 | 1 | 0

2. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Physical and Neurological Examination Findings up to 12 Months
Description: Physical examination assessed: general appearance, dermatological, head and eyes, ears, nose, mouth, and throat, pulmonary, cardiovascular, abdominal, genitourinary (optional), lymphatic, musculoskeletal/extremities. Neurological examination assessed: level of consciousness, mental status, cranial nerve assessment, muscle strength and tone, reflexes, pin prick and vibratory sensation, coordination and gait. Investigator judged clinically significant change from baseline in physical and neurological examination findings.
Time Frame: Baseline up to 12 Months
Population: Safety population included participants who took at least 1 dose of the study medication in the study. Here, "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin: Previous and Current | Placebo-Previous to Pregabalin-Current | Direct Pregabalin
Number analyzed (Participants) | 384 | 210 | 11
Participants
  Physical Examination: number analyzed (Participants) | 369 | 199 | 9
  Physical Examination | 8 | 6 | 0
  Neurological Examination: number analyzed (Participants) | 368 | 199 | 9
  Neurological Examination | 10 | 4 | 2

3. Primary Outcome: Number of Participants Meeting Pre-defined Criteria for Vital Signs Abnormalities
Description: Pre-defined criteria of vital signs abnormalities: maximum (max.) increase or decrease from baseline in sitting/supine systolic blood pressure (SBP) >=30 millimeter of mercury (mmHg); maximum increase or decrease from baseline in sitting/supine diastolic blood pressure (DBP) >=20 mmHg.
Time Frame: Baseline up to 12 months
Population: Safety population included participants who took at least 1 dose of the study medication in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin: Previous and Current | Placebo-Previous to Pregabalin-Current | Direct Pregabalin
Number analyzed (Participants) | 384 | 210 | 11
Participants
  Max. increase from baseline in SBP>=30 mmHg | 9 | 1 | 0
  Max. decrease from baseline in SBP>=30 mmHg | 8 | 5 | 0
  Max. increase from baseline in DBP>=20 mmHg | 34 | 16 | 1
  Max. decrease from baseline in DBP>=20 mmHg | 22 | 6 | 0

4. Primary Outcome: Number of Participants With Tanner Staging Evaluation at Baseline
Description: Tanner stage defines physical measurements of development based on external primary and secondary sex characteristics. Participants were evaluated for pubic hair distribution, breast development (only females) and genital development (only males), with values ranging from stage 1 (pre-pubertal characteristics) to stage 5 (adult or mature characteristics).
Time Frame: Baseline (Day 1)
Population: Analysis population included who took at least 1 dose of the study medication in the study and with age 4 years to less than 17 years. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure and "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin: Previous and Current | Placebo-Previous to Pregabalin-Current | Direct Pregabalin
Number analyzed (Participants) | 213 | 98 | 9
Participants
  Pubic Hair: number analyzed (Participants) | 212 | 98 | 9
  Pubic Hair: Stage 1 | 95 | 44 | 4
  Pubic Hair: Stage 2 | 34 | 17 | 1
  Pubic Hair: Stage 3 | 33 | 16 | 0
  Pubic Hair: Stage 4 | 34 | 15 | 0
  Pubic Hair: Stage 5 | 16 | 6 | 2
  Pubic Hair: Not Done | 0 | 0 | 2
  Pubic Hair: Missing | 0 | 0 | 0
  Breast: number analyzed (Participants) | 122 | 52 | 6
  Breast: Stage 1 | 37 | 18 | 2
  Breast: Stage 2 | 17 | 8 | 1
  Breast: Stage 3 | 15 | 7 | 0
  Breast: Stage 4 | 19 | 7 | 0
  Breast: Stage 5 | 9 | 3 | 2
  Breast: Not Done | 1 | 0 | 1
  Breast: Missing | 24 | 9 | 0
  Genitalia: number analyzed (Participants) | 133 | 64 | 3
  Genitalia: Stage 1 | 50 | 23 | 2
  Genitalia: Stage 2 | 24 | 11 | 0
  Genitalia: Stage 3 | 20 | 10 | 0
  Genitalia: Stage 4 | 13 | 7 | 0
  Genitalia: Stage 5 | 7 | 3 | 0
  Genitalia: Not Done | 0 | 1 | 1
  Genitalia: Missing | 19 | 9 | 0

5. Primary Outcome: Number of Participants With Tanner Staging Evaluation at Month 12
Description: as for outcome 4
Time Frame: Month 12
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin: Previous and Current | Placebo-Previous to Pregabalin-Current | Direct Pregabalin
Number analyzed (Participants) | 186 | 89 | 5
Participants
  Pubic Hair: Stage 1 | 68 | 38 | 2
  Pubic Hair: Stage 2 | 35 | 17 | 1
  Pubic Hair: Stage 3 | 38 | 12 | 0
  Pubic Hair: Stage 4 | 21 | 11 | 0
  Pubic Hair: Stage 5 | 23 | 10 | 1
  Pubic Hair: Not Done | 1 | 1 | 1
  Pubic Hair: Missing | 0 | 0 | 0
  Breast: number analyzed (Participants) | 82 | 37 | 4
  Breast: Stage 1 | 27 | 15 | 2
  Breast: Stage 2 | 17 | 8 | 1
  Breast: Stage 3 | 19 | 5 | 0
  Breast: Stage 4 | 7 | 3 | 0
  Breast: Stage 5 | 12 | 5 | 1
  Breast: Not Done | 0 | 1 | 0
  Breast: Missing | 0 | 0 | 0
  Genitalia: number analyzed (Participants) | 104 | 52 | 1
  Genitalia: Stage 1 | 40 | 19 | 1
  Genitalia: Stage 2 | 22 | 12 | 0
  Genitalia: Stage 3 | 20 | 10 | 0
  Genitalia: Stage 4 | 9 | 5 | 0
  Genitalia: Stage 5 | 13 | 6 | 0
  Genitalia: Not Done | 0 | 0 | 0
  Genitalia: Missing | 0 | 0 | 0

6. Primary Outcome: Number of Participants With >=7 Percent (%) Change From Baseline in Body Weight up to 12 Months
Description: In this outcome measure number of participants with increase and decrease of >=7% in body weight, from baseline up to 12 months are reported.
Time Frame: Baseline up to 12 Months
Population: Safety population included participants who took at least 1 dose of the study medication in the study. Here "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin: Previous and Current | Placebo-Previous to Pregabalin-Current | Direct Pregabalin
Number analyzed (Participants) | 377 | 203 | 9
Participants
  Weight increase from baseline >=7% | 290 | 147 | 8
  Weight decrease from baseline >=7% | 2 | 4 | 0

7. Primary Outcome: Absolute Values for Body Height at Baseline
Time Frame: Baseline
Population: Safety population included participants who took at least 1 dose of the study medication in the study. Here,"Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Pregabalin: Previous and Current | Placebo-Previous to Pregabalin-Current | Direct Pregabalin
Number analyzed (Participants) | 384 | 210 | 11
Centimeters
  Age: 1 Month to <2 Years: number analyzed (Participants) | 37 | 23 | 0
  Age: 1 Month to <2 Years | 74.7 (7.91) | 74.8 (8.24) |
  Age: 2 Years to <4 Years: number analyzed (Participants) | 60 | 42 | 0
  Age: 2 Years to <4 Years | 92.2 (7.13) | 91.0 (8.21) |
  Age: 4 Years to <10 Years: number analyzed (Participants) | 92 | 43 | 4
  Age: 4 Years to <10 Years | 119.3 (15.16) | 118.5 (11.36) | 126.0 (12.60)
  Age: 10 Years to 16 Years: number analyzed (Participants) | 126 | 57 | 7
  Age: 10 Years to 16 Years | 153.5 (14.50) | 154.7 (11.88) | 153.4 (7.06)
  Age: >=17 Years: number analyzed (Participants) | 69 | 45 | 0
  Age: >=17 Years | 170.4 (9.18) | 170.7 (9.99) |

8. Primary Outcome: Absolute Values for Body Height at Month 12
Time Frame: Month 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Pregabalin: Previous and Current | Placebo-Previous to Pregabalin-Current | Direct Pregabalin
Number analyzed (Participants) | 377 | 202 | 9
Centimeters
  Age: 1 Month to <2 Years: number analyzed (Participants) | 36 | 22 | 0
  Age: 1 Month to <2 Years | 84.4 (7.27) | 85.3 (9.01) |
  Age: 2 Years to <4 Years: number analyzed (Participants) | 58 | 39 | 0
  Age: 2 Years to <4 Years | 99.3 (7.90) | 98.1 (8.94) |
  Age: 4 Years to <10 Years: number analyzed (Participants) | 91 | 43 | 3
  Age: 4 Years to <10 Years | 128.2 (15.94) | 126.6 (10.80) | 128.2 (13.08)
  Age: 10 Years to 16 Years: number analyzed (Participants) | 125 | 55 | 6
  Age: 10 Years to 16 Years | 158.1 (13.64) | 160.5 (11.87) | 153.7 (6.58)
  Age: >=17 Years: number analyzed (Participants) | 67 | 43 | 0
  Age: >=17 Years | 170.8 (9.54) | 170.6 (10.14) |

9. Primary Outcome: Number of Participants With Incidence of Laboratory Abnormalities
Description: Criteria for laboratory abnormalities: Hemoglobin (Hgb), hematocrit, red blood cell(RBC) count: <0.8*lower limit of normal(LLN), platelet: <0.5*LLN/greater than (>)1.75*upper limit of normal (ULN), white blood cell (WBC): <0.6*LLN/>1.5*ULN, lymphocyte, neutrophil- absolute/%:<0.8*LLN/>1.2*ULN, basophil, eosinophil, monocyte- absolute/%:>1.2*ULN; total/direct/indirect bilirubin >1.5*ULN, aspartate aminotransferase (AT), alanine AT, gammaglutamyl transferase, alkaline phosphatase:> 3.0*ULN, total protein, albumin: <0.8*LLN/>1.2*ULN; thyroxine, thyroid stimulating hormone <0.8*LLN/>1.2*ULN; cholesterol, triglycerides:> >1.3*ULN; blood urea nitrogen, creatinine:>1.3*ULN; sodium <0.95*LLN/>1.05*ULN, potassium, chloride, calcium: <0.9*LLN or >1.1*ULN; glucose <0.6*LLN/>1.5*ULN, creatine kinase>2.0*ULN; urine (specific gravity <1.003/>1.030, pH <4.5/>8, glucose, ketones, protein: >=1, WBC, RBC:>=20, bacteria >20, hyaline casts/casts >1); prothrombin (PT), PT international ratio>1.1*ULN.
Time Frame: Baseline up to 12 Months
Population: Analysis population included participants who took at least 1 dose of the study medication in the study and were evaluable for laboratory abnormalities.
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin: Previous and Current | Placebo-Previous to Pregabalin-Current | Direct Pregabalin
Number analyzed (Participants) | 374 | 204 | 9
Participants | 297 | 164 | 8

10. Primary Outcome: Number of Participants With Maximum Change From Baseline up to 12 Months in 12-Lead Electrocardiogram (ECG) Parameters
Description: Categories for which data is reported are: 1) maximum (max) PR interval increase from baseline (IFB) (millisecond [msec]) percent change (PctChg) >=25/50%; 2) maximum QRS complex increase from baseline (msec) PctChg>=50%; 3) maximum QTcB interval (Bazett's correction) increase from baseline (msec): change >=30 to <60; change >=60; 4) maximum QTcF interval (Fridericia's correction) increase from baseline (msec): change >=30 to <60; change >=60. 'PctChg>=25/50%': >= 25% increase from baseline when baseline ECG parameter is > 200 msec, and is >= 50% increase from baseline when baseline ECG parameter is non-missing and <=200 msec.
Time Frame: Baseline up to 12 Months
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin: Previous and Current | Placebo-Previous to Pregabalin-Current | Direct Pregabalin
Number analyzed (Participants) | 357 | 194 | 9
Participants
  Max PR interval IFB PctChg >=25/50% | 1 | 0 | 0
  Max QRS complex IFB PctChg >=50% | 0 | 0 | 0
  Max QTcB interval IFB change >=30 - <60 | 29 | 11 | 0
  Max QTcB interval IFB change >=60 | 0 | 0 | 0
  Max QTcF interval IFB change >=30 - <60 | 18 | 9 | 1
  Max QTcF interval IFB change >=60 | 1 | 0 | 0

11. Primary Outcome: 28-Days Seizure Rate at Week 1
Description: 28-days seizure rate was defined as number of seizures per 28-day period. 28-days seizure rate have been reported separately for partial onset seizure and primary generalized tonic clonic seizure. Partial onset seizure: a seizure that starts in one area of the brain. This kind of seizure is brief, lasting seconds to less than 2 minutes. Primary generalized tonic clonic seizure: a seizure that starts in one area of the brain, then spreads to both sides of the brain as a tonic-clonic seizure and usually last 1 to 3 minutes.
Time Frame: Week 1
Population: Safety population included participants who took at least 1 dose of the study medication in the study. Here "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure and "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Seizures Per 28-Days
Arm/Group | Pregabalin: Previous and Current | Placebo-Previous to Pregabalin-Current | Direct Pregabalin
Number analyzed (Participants) | 380 | 209 | 11
Seizures Per 28-Days
  Partial Onset Seizures: number analyzed (Participants) | 270 | 147 | 11
  Partial Onset Seizures | 102.89 (235.73) | 190.45 (1143.83) | 17.83 (32.18)
  Primary Generalized Tonic Clonic Seizures: number analyzed (Participants) | 110 | 62 | 0
  Primary Generalized Tonic Clonic Seizures | 2.07 (2.98) | 2.39 (4.53) |

12. Primary Outcome: 28-Days Seizure Rate at Month 1
Description: as for outcome 11
Time Frame: Month 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Seizures Per 28-Days
Arm/Group | Pregabalin: Previous and Current | Placebo-Previous to Pregabalin-Current | Direct Pregabalin
Number analyzed (Participants) | 378 | 203 | 10
Seizures Per 28-Days
  Partial Onset Seizures: number analyzed (Participants) | 269 | 142 | 10
  Partial Onset Seizures | 96.39 (258.09) | 178.53 (1114.79) | 33.42 (54.21)
  Primary Generalized Tonic Clonic Seizures: number analyzed (Participants) | 109 | 61 | 0
  Primary Generalized Tonic Clonic Seizures | 1.43 (2.16) | 1.66 (2.86) |

13. Primary Outcome: 28-Days Seizure Rate at Month 2
Description: as for outcome 11
Time Frame: Month 2
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Seizures Per 28-Days
Arm/Group | Pregabalin: Previous and Current | Placebo-Previous to Pregabalin-Current | Direct Pregabalin
Number analyzed (Participants) | 373 | 193 | 8
Seizures Per 28-Days
  Partial Onset Seizures: number analyzed (Participants) | 263 | 135 | 8
  Partial Onset Seizures | 79.33 (196.31) | 89.09 (579.42) | 22.16 (46.70)
  Primary Generalized Tonic Clonic Seizures: number analyzed (Participants) | 110 | 58 | 0
  Primary Generalized Tonic Clonic Seizures | 1.27 (1.80) | 1.36 (2.63) |

14. Primary Outcome: 28-Days Seizure Rate at Month 4
Description: as for outcome 11
Time Frame: Month 4
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Seizures Per 28-Days
Arm/Group | Pregabalin: Previous and Current | Placebo-Previous to Pregabalin-Current | Direct Pregabalin
Number analyzed (Participants) | 352 | 185 | 6
Seizures Per 28-Days
  Partial Onset Seizures: number analyzed (Participants) | 247 | 131 | 6
  Partial Onset Seizures | 67.32 (190.44) | 58.33 (320.32) | 15.45 (25.23)
  Primary Generalized Tonic Clonic Seizures: number analyzed (Participants) | 105 | 54 | 0
  Primary Generalized Tonic Clonic Seizures | 1.09 (1.88) | 0.72 (0.91) |

15. Primary Outcome: 28-Days Seizure Rate at Month 6
Description: as for outcome 11
Time Frame: Month 6
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Seizures Per 28-Days
Arm/Group | Pregabalin: Previous and Current | Placebo-Previous to Pregabalin-Current | Direct Pregabalin
Number analyzed (Participants) | 330 | 175 | 6
Seizures Per 28-Days
  Partial Onset Seizures: number analyzed (Participants) | 237 | 124 | 6
  Partial Onset Seizures | 50.18 (125.26) | 51.10 (212.59) | 4.25 (6.06)
  Primary Generalized Tonic Clonic Seizures: number analyzed (Participants) | 93 | 51 | 0
  Primary Generalized Tonic Clonic Seizures | 1.02 (1.61) | 0.79 (1.21) |

16. Primary Outcome: 28-Days Seizure Rate at Month 9
Description: as for outcome 11
Time Frame: Month 9
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Seizures Per 28-Days
Arm/Group | Pregabalin: Previous and Current | Placebo-Previous to Pregabalin-Current | Direct Pregabalin
Number analyzed (Participants) | 310 | 164 | 6
Seizures Per 28-Days
  Partial Onset Seizures: number analyzed (Participants) | 225 | 121 | 6
  Partial Onset Seizures | 38.17 (87.75) | 43.13 (141.96) | 3.00 (3.93)
  Primary Generalized Tonic Clonic Seizures: number analyzed (Participants) | 85 | 43 | 0
  Primary Generalized Tonic Clonic Seizures | 0.96 (1.69) | 0.62 (0.99) |

17. Secondary Outcome: Number of Participants With Suicidal Ideation as Per Columbia Suicide Severity Rating Scale (C-SSRS) Mapped to Columbia Classification Algorithm of Suicide Assessment (C-CASA)
Description: Number of participants with C-CASA code 4 are reported. C-SSRS responses mapping to C-CASA suicidal ideation code 4 are as follows: "Yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with any methods (not plan) without intent to act", "active suicidal ideation with some intent to act, without specific plan", "active suicidal ideation with some intent to act, without specific plan".
Time Frame: Baseline (Day 1), Post-baseline on Day 1 up to 12 Months
Population: Analysis population included participants who took at least 1 dose of the study medication in the study and with age >=6 years. Here, "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin: Previous and Current | Placebo-Previous to Pregabalin-Current | Direct Pregabalin
Number analyzed (Participants) | 258 | 134 | 10
Participants
  Baseline: number analyzed (Participants) | 254 | 132 | 10
  Baseline | 3 | 2 | 1
  Post-baseline on Day 1 up to 12 Months: number analyzed (Participants) | 257 | 134 | 10
  Post-baseline on Day 1 up to 12 Months | 3 | 2 | 0

18. Secondary Outcome: Number of Participants With Suicidal Behavior as Per Columbia Suicide Severity Rating Scale (C-SSRS) Mapped to Columbia Classification Algorithm of Suicide Assessment (C-CASA)
Description: Number of participants with C-CASA code 1 or 2 or 3 are reported. C-SSRS responses mapping to C-CASA suicidal behavior codes 1, 2, or 3 are as follows: (1) completed suicide; (2) suicide attempt (response of "Yes" on "actual attempt"); (3) preparatory acts toward imminent suicidal behavior ("Yes" on "aborted attempt", "interrupted attempt", "preparatory acts or behavior").
Time Frame: Baseline (Day 1), Post-baseline up to 12 Months
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin: Previous and Current | Placebo-Previous to Pregabalin-Current | Direct Pregabalin
Number analyzed (Participants) | 258 | 134 | 10
Participants
  Baseline: number analyzed (Participants) | 254 | 132 | 10
  Baseline | 1 | 1 | 0
  Post-baseline on Day 1 up to 12 Months: number analyzed (Participants) | 257 | 134 | 10
  Post-baseline on Day 1 up to 12 Months | 2 | 0 | 0

19. Secondary Outcome: Number of Participants as Per Reliable Change Index (RCI) Category for Cogstate Detection Task
Description: CogState brief battery consisted of 2 tasks- detection and pediatric identification task using a laptop computer with external response buttons. Prior tasks, participants were briefed rules, given an interactive demonstration and a sufficient number of practice trials. For each task, participant responded "yes" using a response button with dominant hand. Participants had to "respond as fast and as accurately as possible." Detection task: measured simple reaction time to assess psychomotor function. Participant pressed a "YES" response key as soon as they detected an event (ie, a card turning face up presented in the center of the computer screen). A participant's RCI was calculated by dividing the change from individual baseline score by ([square root 2] times WSD), where WSD is within-subject standard deviation from Cogstate detection task normative data. Improvement in cognition when RCI <=-1.65, decline in cognition when RCI =>1.65.
Time Frame: Month 12
Population: Analysis population included participants who took at least 1 dose of the study medication in the study and were evaluable for cognitive testing. Here "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin: Previous and Current | Placebo-Previous to Pregabalin-Current | Direct Pregabalin
Number analyzed (Participants) | 97 | 51 | 7
Participants
  Improvement (RCI <= -1.65) | 21 | 8 | 2
  Decline (RCI =>1.65) | 13 | 6 | 1

20. Secondary Outcome: Number of Participants as Per Reliable Change Index Category for Cogstate Pediatric Identification Task
Description: CogState brief battery consisted of 2 tasks-detection and pediatric identification task using a laptop computer with external response buttons. Prior tasks, participants were briefed rules, given an interactive demonstration and a sufficient number of practice trials. For each task, participant responded "yes" using a response button with dominant hand. Participants had to "respond as fast and as accurately as possible." Pediatric identification task: measured choice reaction time to assess visual attention. An event (a card turning face up) occurred in center of computer screen and participant decided if event met a predefined and unchanging criterion (is the color of the card black?); answered "YES" if criterion was met. A participant's RCI was calculated by dividing the change from individual baseline score by ([square root 2] times WSD),WSD=within-subject standard deviation from Cogstate task normative data. Improvement in cognition: RCI <=-1.65, decline in cognition: RCI =>1.65.
Time Frame: Month 12
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin: Previous and Current | Placebo-Previous to Pregabalin-Current | Direct Pregabalin
Number analyzed (Participants) | 96 | 50 | 7
Participants
  Improvement (RCI <=-1.65) | 17 | 9 | 2
  Decline (RCI =>1.65) | 16 | 6 | 2

21. Primary Outcome: 28-Days Seizure Rate at Month 12/Early Termination
Description: as for outcome 11
Time Frame: Month 12/Early Termination
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Seizures Per 28-Days
Arm/Group | Pregabalin: Previous and Current | Placebo-Previous to Pregabalin-Current | Direct Pregabalin
Number analyzed (Participants) | 374 | 206 | 8
Seizures Per 28-Days
  Partial Onset Seizures: number analyzed (Participants) | 266 | 146 | 8
  Partial Onset Seizures | 56.04 (147.20) | 117.88 (896.40) | 11.08 (16.55)
  Primary Generalized Tonic Clonic Seizures: number analyzed (Participants) | 108 | 60 | 0
  Primary Generalized Tonic Clonic Seizures | 1.02 (1.71) | 1.33 (3.20) |

ADVERSE EVENTS:
Time Frame: Baseline up to 13 Months
Description: Same event may appear as adverse event (AE) and serious AE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as nonserious in another participant or 1 participant may have experienced both serious and nonserious event during study. Safety population was evaluated.
Arm/Group | Pregabalin: Previous and Current | Placebo-Previous to Pregabalin-Current | Direct Pregabalin
All-Cause Mortality (participants affected / at risk) | 3/384 | 4/210 | 0/11
Serious Adverse Events (participants affected / at risk) | 53/384 | 23/210 | 1/11
Other Adverse Events (participants affected / at risk) | 186/384 | 103/210 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin: Previous and Current (N=384) | Placebo-Previous to Pregabalin-Current (N=210) | Direct Pregabalin (N=11)
Deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 0
Cyanosis (Cardiac disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Gingival hypertrophy (Gastrointestinal disorders) | 0 | 1 | 0
Saliva discolouration (Gastrointestinal disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 3 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Dengue fever (Infections and infestations) | 1 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 3 | 0
Giardiasis (Infections and infestations) | 0 | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0
Pharyngotonsillitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 17 | 6 | 0
Respiratory tract chlamydial infection (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Systemic viral infection (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0
Viral infection (Infections and infestations) | 2 | 0 | 0
Brain herniation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 2 | 0 | 0
Epiphyseal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Unintentional medical device removal (Injury, poisoning and procedural complications) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Periostitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Brain oedema (Nervous system disorders) | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 2 | 0
Partial seizures (Nervous system disorders) | 3 | 0 | 0
Postictal state (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 8 | 6 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0
Status epilepticus (Nervous system disorders) | 2 | 0 | 0
Device dislocation (Product Issues) | 1 | 0 | 0
Device occlusion (Product Issues) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Emotional disorder (Psychiatric disorders) | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 2 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Physical abuse (Social circumstances) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin: Previous and Current (N=384) | Placebo-Previous to Pregabalin-Current (N=210) | Direct Pregabalin (N=11)
Abdominal pain upper (Gastrointestinal disorders) | 4 | 1 | 2
Constipation (Gastrointestinal disorders) | 10 | 4 | 1
Diarrhoea (Gastrointestinal disorders) | 20 | 9 | 1
Vomiting (Gastrointestinal disorders) | 15 | 11 | 2
Fatigue (General disorders) | 8 | 2 | 1
Pyrexia (General disorders) | 54 | 22 | 1
Lyme disease (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 26 | 12 | 0
Pneumonia (Infections and infestations) | 13 | 12 | 0
Sinusitis (Infections and infestations) | 2 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 60 | 30 | 0
Viral infection (Infections and infestations) | 15 | 11 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 6 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood triglycerides increased (Investigations) | 1 | 3 | 1
Platelet count abnormal (Investigations) | 0 | 0 | 1
Red blood cell count abnormal (Investigations) | 0 | 0 | 1
Weight increased (Investigations) | 28 | 12 | 2
White blood cell count abnormal (Investigations) | 0 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 10 | 9 | 2
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 3 | 2 | 1
Dizziness (Nervous system disorders) | 19 | 10 | 1
Dysdiadochokinesis (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 24 | 8 | 4
Lethargy (Nervous system disorders) | 1 | 1 | 1
Psychomotor hyperactivity (Nervous system disorders) | 4 | 2 | 1
Resting tremor (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 22 | 12 | 1
Somnolence (Nervous system disorders) | 26 | 27 | 1
Abnormal behaviour (Psychiatric disorders) | 1 | 0 | 1
Aggression (Psychiatric disorders) | 5 | 2 | 1
Behaviour disorder (Psychiatric disorders) | 2 | 2 | 1
Mood altered (Psychiatric disorders) | 1 | 0 | 1
Mood swings (Psychiatric disorders) | 0 | 0 | 1
Staring (Psychiatric disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 23 | 14 | 0
Rash (Skin and subcutaneous tissue disorders) | 9 | 3 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
1 death occurred in reporting arm "Placebo-Previous to Pregabalin-Current" after participant completed the study and is captured in All-cause mortality section.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2014-05-07): https://cdn.clinicaltrials.gov/large-docs/06/NCT01463306/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-03): https://cdn.clinicaltrials.gov/large-docs/06/NCT01463306/SAP_001.pdf